CLINICAL TRIAL: NCT06083467
Title: Center Without Walls for Imaging Proteinopathies With PET (CW2IP2): Imaging and Diagnostic Assessments
Brief Title: CW2IP2: Imaging and Diagnostic Assessments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ilya Nasrallah, Principal Investigator, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 852796
Record Dates: First submitted 2023-07-25; First posted 2023-10-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Tauopathies
Keywords: Amyloid PET; Movement disorders
MeSH Terms: conditions — Tauopathies; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Diagnostic Assessments (Other): Subjects may receive a brain MRI and neurological exam with diagnostic assessments.
  Interventions: Diagnostic Test: Brain MRI Scan; Behavioral: Neurologic exam

INTERVENTIONS:
Diagnostic Test: Brain MRI Scan — MRI scan of the brain
Behavioral: Neurologic exam — Neurologic exam and assessments, including video interview

SUMMARY:
This current protocol will provide the key data to help determine the specificity of our to-be-developed radiotracers by implementing a multi-site diagnostic assessment core and PET imaging of A-beta amyloid (may be completed at some sites as part of another protocol) that is commonly deposited in the brains of people with Parkinson's Disease (PD), Multiple System Atrophy (MSA), Progressive Supranuclear Palsy (PSP) or Frontotemporal Dementia (FTD) as well as healthy controls. This multicenter U19 grant is centered at U Pennsylvania (U Penn) (PI: Robert Mach) in collaboration with U Pittsburgh (Pitt), Yale University, U of California at San Francisco (UCSF) and Washington University in St. Louis (WU). U Penn will act as the single IRB of Record (sIRB) for this multi-center project and subjects will be recruited from all sites.

DETAILED DESCRIPTION:
This current protocol will provide the key data to help determine the specificity of our to-be-developed radiotracers by implementing a multi-site diagnostic assessment core to be compared with new radiotracer scans for 4RTau and Alphasynuclein which are compounds in the brains of people with Parkinson's Disease (PD), Multiple System Atrophy (MSA), Progressive Supranuclear Palsy (PSP) or Frontotemporal Dementia (FTD) as well as healthy controls. This multicenter U19 grant is centered at U Pennsylvania (U Penn) (PI: Robert Mach) in collaboration with U Pittsburgh (Pitt), Yale University, U of California at San Francisco (UCSF) and Washington University in St. Louis (WU). U Penn will act as the single IRB of Record (sIRB) for this multi-center project and subjects will be recruited from all sites. Sites will have local Radiation Research Safety Committee or Radioactive Drug Research Committee oversight over radiation safety related issues specific to the A-beta amyloid radiotracer used at that site (Florbetaben (18F) or 11C-PiB), if the site chooses to include A-beta amyloid PET imaging. Some sites may participate in this diagnostic assessment study without the PET/CT imaging if that data is collected as part of other studies conducted at the site.

The investigators will recruit up to 10 people with PD, 10 healthy controls, 10 with MSA, 10 with PSP and 14 with FTD (4 of these FTD participants are expected tau-negative FTD controls and 10 are expected tau-positive).

Key components of the multi-site diagnostic core will provide the infrastructure for these human imaging studies including regulatory activities (with a sIRB, at Penn); consistency of diagnostic criteria and clinical evaluations (with clinical consensus diagnosis of all participants); common calibration of PET scanners; model consents and protocols; and collection and distribution of clinical and imaging data.

Subjects will be required to have a brain MRI performed within 12 months of study enrollment. If the subject has not had a brain MRI that is deemed acceptable for use for this study by an investigator, they will be asked to undergo a research brain MRI after they have consented for this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants: Patients in all cohorts will range from 40 to 85 yrs and will be both male and female.
* Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures. Participants who are deemed unable to provide informed consent must have a designated Legally Authorized Representative(LAR) present for consent and a Study Partner to accompany them to study visits. The LAR and the Study Partner may be the same person.
* Clinical diagnoses for each cohort will be determined by consensus committee for diagnostic agreement (PD, MSA, PSP, FTD or Healthy control)

Exclusion Criteria:

* Females who are pregnant or breast feeding at the time of screening will be excluded
* Forms of parkinsonism other than PD, PSP and MSA as defined above
* Major psychiatric disorder (e.g. schizophrenia or bipolar disorder)
* History of significant or ongoing alcohol abuse or substance abuse or dependence based on medical record review or self-reported
* Contraindications or Inability to tolerate imaging, arterial line or IV placement or blood draw procedures in the opinion of an investigator or treating physician
* Implanted medical device or other contraindication to MRI
* Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician or investigator to be a condition that could compromise participant safety or successful participation in the study
* Refusal to consent to brain donation (except for HC cohort). All non-HC participants must agree to postmortem brain donation..

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Disease diagnosis | 8 weeks
  The primary outcome is a diagnosis classification of a neurodegenerative disease. Participants will be referred based on a clinical evaluation suggesting possible Parkinson Disease, Progressive Supranuclear Palsy, Multiple System Atrophy, Frontotemporal Lobar Degeneration, or other neurodegenerative disease or as a likely healthy control. Participants will have cognitive testing, physical examination, imaging studies, and record review, which will be used to determine the probable diagnosis. If no probable diagnosis is achieved, the outcome would be an uncertain diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A request to utilize de-identified data will be reviewed by the Clinical Core Oversight Committee (CCOC). Each investigator using data is required to sign a Use Agreement form that stipulates the following:
  * Data received will only be used for the purposes stated in the study design.
  * Received data will not be distributed to others (apart from collaborators named in the study).
  * The investigator will not attempt to directly or indirectly identify participants.
  * Results will be made available to the research community in a timely manner and acknowledge CW2IP2.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Screening data including neurologic assessments, brain MRI and Amyloid PET results shared when collected. Clinical study report after completion of the study.